CLINICAL TRIAL: NCT05643742
Title: A Phase 1/2, Open-Label, Multicenter, Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Anti-CD19 Allogeneic CRISPR-Cas9-Engineered T Cells (CTX112) in Subjects With Relapsed or Refractory B Cell Malignancies
Brief Title: A Safety and Efficacy Study Evaluating CTX112 in Subjects With Relapsed or Refractory B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-006
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: B-cell Lymphoma; Non-Hodgkin Lymphoma; B-cell Malignancy; Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL); Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Large B-cell Lymphoma
Keywords: CAR T; Non-Hodgkin Lymphoma (NHL); Lymphoma; Allogeneic
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX112 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX112

INTERVENTIONS:
Biological: CTX112 — CTX112 (CD19-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components)

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study evaluating the safety and efficacy of CTX112™ in subjects with relapsed or refractory B-cell malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 1/2 study of CTX112 in subjects with relapsed/refractory B cell malignancies. CTX112 is an is allogeneic CD19-directed chimeric antigen receptor (CAR) T cell immunotherapy comprised of allogeneic T cells that are genetically modified ex vivo using CRISPR-Cas9 (clustered regularly interspaced short palindromic repeats/ CRISPR associated protein 9) gene editing components (single guide RNA and Cas9 nuclease).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years.
2. Refractory or relapsed B cell malignancy.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Adequate renal, liver, cardiac and pulmonary organ function.
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX112 infusion.

Key Exclusion Criteria:

1. Prior allogeneic hematopoietic stem cell transplant (HSCT).
2. Active or history of central nervous system (CNS) involvement by malignancy.
3. History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
4. Presence of bacterial, viral, or fungal infection that is uncontrolled or requires IV anti-infectives.
5. Active HIV, hepatitis B virus or hepatitis C virus infection.
6. Previous or concurrent malignancy in the last 3 years (with the exception of non-melanoma skin cancer and other cancers deemed by the investigator and medical monitor to be of low likelihood for recurrence).
7. Concurrent systemic treatment with an anticancer biologic (e.g., monoclonal antibody) within 30 days prior to CTX112 infusion or with a nonbiological anticancer drug within 14 days prior to CTX112 infusion.
8. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
9. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation): Incidence of adverse events, defined as dose-limiting toxicities | From CTX112 infusion up to 28 days post-infusion
Phase 2 (Cohort Expansion): Objective response rate | From CTX112 infusion up to 60 months post-infusion

SECONDARY OUTCOMES:
Duration of Response | From date of first objective response of complete response (CR)/partial response (PR) until date of disease progression or death due to any cause, assessed up to 60 months
  Duration of Response (DOR) will only be reported for subjects who have had CR/PR events
Duration of Clinical Benefit (DOCB) | From date of first objective response of CR/PR until the relapse or death that followed the last response, assessed up to 60 months
Progression Free Survival | From date of CTX112 infusion until date of disease progression or death due to any cause, assessed up to 60 months
Overall Survival | From date of CTX112 infusion until date of death due to any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Allen, M.Sc., Study Director — CRISPR Therapeutics
Locations (7):
- United States (4):
  - University of Kansas, Westwood, Kansas
  - Washington University, St Louis, Missouri
  - SCRI, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Royal Prince Alfred, Camperdown, New South Wales
  - Alfred Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No